CLINICAL TRIAL: NCT04546698
Title: 5-HTSEP: Serotonin 5-HT7 Receptor Implication in the Inflammatory Mechanisms in Multiple Sclerosis
Brief Title: 5-HT7 Receptor Implication in Inflammatory Mechanisms in Multiple Sclerosis
Acronym: 5-HTSEP
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Régional d'Orléans (Other)
Collaborators: National Scientific Research Centre (Unknown)
Responsible Party: Sponsor
Other Study IDs: CHRO-2020-01
Record Dates: First submitted 2020-08-31; First posted 2020-09-14 (Actual); Last update posted 2022-02-17 (Actual); Status verified 2022-02

CONDITIONS: Multiple Sclerosis, Acute Relapsing; Multiple Sclerosis
Keywords: Multiple sclerosis; serotonin; 5-HT7 receptor; inflammation; lymphocytes; cytokines
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis; Inflammation | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — one sampling to assess nvestigate the expression modulation of 5-HT7 receptor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Multiple Sclerosis patients with an acute relapse: Multiple Sclerosis diagnosed according to Mc Donald's criteria with an acute relapse
  Interventions: Other: blood sampling
- Multiple sclerosis pataients treated with Natalizumab: Multiple Sclerosis patients diagnosed according to Mc Donald's criteria and treated with Natalizumab since 6 cures
  Interventions: Other: blood sampling
- Healthy people
  Interventions: Other: blood sampling

INTERVENTIONS:
Other: blood sampling — Analyse of expression modulation of 5-HT7 receptor in correlation with the immunological context, in 3 differents groups : 2 with multiple sclerosis patients, one healthy volunteers group

SUMMARY:
Multiple Sclerosis is a chronic autoimmune disease associated with inflammatory response harmful for the Central Nervous System. Immunological imbalance is involved with Th1 and Th17 cells in correlation with a disturbance of regulators mechanisms as Treg cells. Despite years of research, the mechanisms involved remain unclear.

Serotonin (5-HT) seems to be a therapeutic target to treat multiple sclerosis. Indeed, several studies have shown the anti-inflammatory potential of this neurotransmitter and also its vulnerability in inflammatory context. Moreover, a recent study has shown that 5-HT can reduced CD4 T cells proliferation and pro-inflammatory cytokines released in vitro.

5-HT protector effects have also demonstrated in Experimental Autoimmune Encephalomyelitis mouse model (EAE) with an inflammatory response reduction and also a decreased of spinal cord lesions.

The latest receptor discovered, the 5-HT7 receptor, has been identify as a promise target to treat neurological disorders associated with inflammatory context. Present in humans and mice, this receptor spreads on the surface of a large number of cells, such as T-lymphocytes, macrophages, dendritic cells and also neurons, astrocytes and microglia.

Given the importance of the positive cells for 5-HT7 receptor, in the inflammatory context observed in multiple sclerosis, The investigator propose to study the receptor expression in blood samples from multiple sclerosis patient.

DETAILED DESCRIPTION:
The expression modulation of 5-HT7 receptor will be investigate in correlation with the immunological context, in different group of MS patients:

* Group 1: MS patients with an acute relapse
* Group 2: MS stable patients treated with Natalizumab
* Group 3: Healthy people (from Etablissement Français du Sang)

  1. 5-HT7 receptor expression evaluation on circulating leukocyte cells Each group presents a different inflammatory context. The investigator wish to determine the immunological context influence on the 5-HT7 receptor expression and which cells express it. To analyze the 5-HT7 expression on circulating leukocyte cells, The investigator will perform flow cytometry studies from the whole blood of the three groups mentioned above. In a first step, the investigator will analyze the overall rate of 5-HT7 circulating positive cells by the use of an antibody against 5-HT7 receptor whose specificity was validated in our research team. In a second step, the investigator will precise which cell type, among the lymphocytes implicated in the MS pathology, express the 5-HT7 receptor. The investigator will use antibodies against each population t helper cell: Th1 , Th2, Th17 and Treg. The investigator will also perform immunostaining on Cytospin (thin layer of blood cells on coverslips) to visualize co-labeling and confirm the results of flow cytometry.
  2. Correlation between 5-HT7 receptor expression and mRNA quantity In addition, a correlation has been shown between an increase of 5-HT7 positive cells and an mRNA quantity up regulated. For the three groups, the investigator will determine the 5-HT7 mRNA quantity on circulating leukocyte cells. In a first step, the investigator will check correlation between the 5-HT7 receptor expression rate and the mRNA quantity on circulating leukocyte cells, using quantitative Polymerase Chain Reaction (qPCR). In a second step, the investigator will perform cell sorting to isolate Th1, Th2, Th17 and Treg cells and specifically extract 5-HT7 mRNA. In this way, the investigator can address the 5-HT7 receptor role on one or more specific cell types on the MS.
  3. 5-HT7 receptor modulation according to the immunological context In order to understand the 5-HT7 receptor potential role on immune response moderation, the investigator will identify the immune context by ELISA dosage from serum samples. The investigator will investigate on pro-inflammatory markers like IL1b, IFNg, IL17 and anti-inflammatory markers like IL10 and IL4. These results will be correlated with the previous results concerning the 5-HT7 receptor expression/quantity for each patient groups.
  4. 5-HT7 receptor role on lymphocyte functions in vitro From blood samples of the three groups mentioned above, the investigator will isolate peripheral blood mononuclear cells (PBMC) in vitro, to evaluate the 5-HT7 receptor role on their function to produce and release cytokines. The investigator will stimulate PBMC with one or more 5-HT7 ligands, and will perform ELISA dosage from supernatant with pro-inflammatory markers like IL1b, IFNg, IL17 and anti-inflammatory markers like IL10 and IL4. The cell immunolabelling will be perform to visualize 5-HT7 receptor on the cell surface.
  5. Identification of 5-HT7 receptor isoforms There are three forms of 5-HT7 receptor (5-HT7a, 5-HT7b, 5-HT7d). However, no difference has yet been described for their pharmacological function. The investigator propose to identify these different isoforms by qPCR. As previously described, in a first step, on circulating leukocyte cells and in a second step, after cell sorting to isolate Th1, Th2, Th17 and Treg cells.

ELIGIBILITY:
Inclusion Criteria:

* Man and Woman
* 18 to 50 years old
* Multiple Sclerosis diagnosed according to Mc Donald's criteria (Thompson et al. 2018)
* With an acute relapse (group 1)
* Stable with Natalizumab treatment (group 2), minimum 6 Natalizumab cures
* Healthy Volunteers (group 3)

Exclusion Criteria:

* without social security
* HIV positive serology
* infectious status in the past month
* corticosteroid therapy in the past month
* dementia
* pregnant or breastfeeding woman
* previous participation in the study
* under judicial protection
* non-cooperating patient

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Man and Woman 18 to 50 years old
Sampling Method: Non-Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2020-09-07 (Actual); Primary Completion 2021-07-19 (Actual); Study Completion 2021-07-19 (Actual)

PRIMARY OUTCOMES:
5HT7 Serotonin receptor expression on circulating leukocyte cells | Baseline
  To analyze the 5-HT7 expression on circulating leukocyte cells, we will perform flow cytometry studies from the whole blood of the three groups mentioned above. In a first step, we will analyze the overall rate of 5-HT7 circulating positive cells by the use of an antibody against 5-HT7 receptor whose specificity was validated in our research team. In a second step, we will precise which cell type, among the lymphocytes implicated in the MS pathology, express the 5-HT7 receptor. We will use antibodies against each population: Thelper 1 cell, Thelper 2 cell, Thelper 17 cell and Treg. We will also perform immunostaining on Cytospin (thin layer of blood cells on coverslips) to visualize co-labeling and confirm the results of flow cytometry.
5-HT7 Serotonin receptor mRNA quantity | Baseline
  For the three groups, we will determine the 5-HT7 mRNA quantity on circulating leukocyte cells. In a first step, we will check correlation between the 5-HT7 receptor expression rate and the mRNA quantity on circulating leukocyte cells, using quantitative Polymerase Chain Reaction (qPCR). In a second step, we will perform cell sorting to isolate Thelper 1 cell, Thelper 2 cell , Thelper 17 cell and Treg cells and specifically extract 5-HT7 mRNA.
Immunological context on blood samples | Baseline
  We will identify the immune context by ELISA dosage from serum samples. We will investigate on pro-inflammatory markers like Interleukin 1b, IFNg, IL17 and anti-inflammatory markers like Interleukin 10 and Interluekin 4.
5-HT7 receptor role on lymphocyte functions in vitro | Baseline
  From blood samples of the three groups mentioned above, we will isolate peripheral blood mononuclear cells (PBMC) in vitro, to evaluate the 5-HT7 receptor role on their function to produce and release cytokines. We will stimulate PBMC with one or more 5-HT7 ligands, and we will perform ELISA dosage from supernatant with pro-inflammatory markers like IL1b, IFNg, IL17 and anti-inflammatory markers like IL10 and IL4. The cell immunolabelling will be perform to visualize 5-HT7 receptor on the cell surface.
5-HT7 receptor isoforms 5-HT7 receptor isoforms | Baseline
  There are three forms of 5-HT7 receptor (5-HT7a, 5-HT7b, 5-HT7d). We propose to identify these different isoforms by qPCR. As previously described, in a first step, on circulating leukocyte cells and in a second step, after cell sorting to isolate Th1, Th2, Th17 and Treg cells.

CONTACTS AND LOCATIONS:
Overall Officials: Maud PALLIX, MD, Principal Investigator — CHR ORLEANS
Locations (1):
- CHR Orléans, Orléans, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Thompson AJ, Banwell BL, Barkhof F, Carroll WM, Coetzee T, Comi G, Correale J, Fazekas F, Filippi M, Freedman MS, Fujihara K, Galetta SL, Hartung HP, Kappos L, Lublin FD, Marrie RA, Miller AE, Miller DH, Montalban X, Mowry EM, Sorensen PS, Tintore M, Traboulsee AL, Trojano M, Uitdehaag BMJ, Vukusic S, Waubant E, Weinshenker BG, Reingold SC, Cohen JA. Diagnosis of multiple sclerosis: 2017 revisions of the McDonald criteria. Lancet Neurol. 2018 Feb;17(2):162-173. doi: 10.1016/S1474-4422(17)30470-2. Epub 2017 Dec 21. PMID 29275977
- [Result] Sacramento PM, Monteiro C, Dias ASO, Kasahara TM, Ferreira TB, Hygino J, Wing AC, Andrade RM, Rueda F, Sales MC, Vasconcelos CC, Bento CAM. Serotonin decreases the production of Th1/Th17 cytokines and elevates the frequency of regulatory CD4+ T-cell subsets in multiple sclerosis patients. Eur J Immunol. 2018 Aug;48(8):1376-1388. doi: 10.1002/eji.201847525. Epub 2018 Jun 6. PMID 29719048
- [Result] Yuan XQ, Qiu G, Liu XJ, Liu S, Wu Y, Wang X, Lu T. Fluoxetine promotes remission in acute experimental autoimmune encephalomyelitis in rats. Neuroimmunomodulation. 2012;19(4):201-8. doi: 10.1159/000334095. Epub 2012 Mar 21. PMID 22441536
- [Result] Quintero-Villegas A, Valdes-Ferrer SI. Role of 5-HT7 receptors in the immune system in health and disease. Mol Med. 2019 Dec 31;26(1):2. doi: 10.1186/s10020-019-0126-x. PMID 31892309